CLINICAL TRIAL: NCT06844630
Title: Comparison of Postoperative Analgesic Efficacy Between the Interscalene Block and Infraspinatus-Teres Minor Interfascial Blocks in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Interscalene vs Infraspinatus-teres Minor (ITM) Interfascial Block in Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kadem Koc (Other)
Responsible Party: Sponsor-Investigator, Kadem Koc, Research Fellow, Samsun University
Organization: Samsun University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SamsunOm
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain; Pain, Postoperative; Surgical Procedure, Unspecified
Keywords: arthroscopic shoulder surgery; postoperative pain; interscalene brachial plexus block; infraspinatus-teres minor interfascial block
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Block (Experimental): Patients randomized to receive interscalene block
  Interventions: Other: Preoperative block application (İntersclane Block)
- Infraspinatus-teres minor (ITM) interfascial block (Experimental): Patients randomized to receive Infraspinatus-teres minor (ITM) interfascial block
  Interventions: Other: Preoperative block application (Infraspinatus-teres minor interfascial block)

INTERVENTIONS:
Other: Preoperative block application (İntersclane Block) — Before surgery, patients will receive a unilateral interscalene block under ultrasound guidance.
  Arms: Interscalene Block
Other: Preoperative block application (Infraspinatus-teres minor interfascial block) — Before surgery, patients will receive a unilateral infraspinatus-teres minor interfascial block under ultrasound guidance.
  Arms: Infraspinatus-teres minor (ITM) interfascial block

SUMMARY:
Postoperative pain is important following arthroscopic shoulder surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay.Ultrasound (US)-guided brachial plexus blocks such as interscalen and supraclavicular block are usually performed. Interscalene brachial plexus block is one of the most preferred techniques among these.

Due to the phrenic nerve paralysis frequently seen in interscalene block, alternative diaphragm-sparing block techniques have emerged over time. One of these is the Infraspinatus teres minor interfascial block. Infraspinatus teres minor interfascial block can block both the suprascapular nerve and the axillary nerve, which are effective in the innervation of the shoulder, with a single-point injection.

The main aim of our study was to show that there is no difference between interscalene block and infraspinatus-teres-minor interfascial block in terms of their effects on postoperative analgesia in patients undergoing arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II-III
* Scheduled for arthroscopic shoulder surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis
* receiving anticoagulant treatment
* infection of the skin at the site of the needle puncture
* pregnancy or lactation
* patients who do not accept the procedure
* Allergy to local anesthetics
* Chronic pain syndromes requiring opioid intake

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
24 hours opioid consumption | Time Frame: up to 24 hours
  morphine consumptions via patient controlled analgesia device for both group will be recorded

SECONDARY OUTCOMES:
Sensory and Motor block score | 30 minutes post injection
  Sensorimotor block assessed every 5 minutes until 30 minutes using a 8-point composite. Block level will be evaluated between 0-8 points score
Numeric rating scale for postoperative pain intensity | up to 24 hours (Will be evaluated at 1, 3, 6, 12, 18, 24 hours)
  Evaluated with a Numerical rating scale (NRS) from 0 to 10. (0=no pain; 10=worst imaginable pain)
Quality of Recovery - 15 score | Postoperative 24th hour
  The impact of surgical and anesthetic interventions on perioperative quality of life and ability to resume routine life activities will be assessed using the Quality of Recovery (QoR) tool. Each question is scored between 0 and 10. The survey result varies between 0-150 points based on the answers given by the patients. Higher scores indicate better recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SH, Yeo IS, Jang J, Jung HE, Chun YM, Yang HM. Infraspinatus-teres minor (ITM) interfascial block: a novel approach for combined suprascapular and axillary nerve block. Reg Anesth Pain Med. 2024 Jan 11;49(1):67-72. doi: 10.1136/rapm-2023-104738. PMID 37491150
- [Background] Aliste J, Bravo D, Layera S, Fernandez D, Jara A, Maccioni C, Infante C, Finlayson RJ, Tran DQ. Randomized comparison between interscalene and costoclavicular blocks for arthroscopic shoulder surgery. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100055. doi: 10.1136/rapm-2018-100055. Online ahead of print. PMID 30635497
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714